CLINICAL TRIAL: NCT01163318
Title: Special Investigation (Long-term Treatment in Patients With Rheumatoid Arthritis)
Brief Title: Special Investigation of Humira® (Adalimumab) on Long-term Treatment in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-070
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adalimumab 40 mg/0.8 mL syringe for subcutaneous injection: Participants with rheumatoid arthritis who received adalimumab, per approved label

SUMMARY:
The purpose of this study was to collect data on the incidence of adverse drug reactions, infections and malignant tumors, as well as factors that might affect the safety and effectiveness of Humira® (adalimumab; 40mg/0.8 mL) in Japanese participants who received the drug for the treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic autoimmune disease which requires long-term treatment. Due to the need of long-term safety data in Japanese participants and to fulfil the conditions of approval of adalimumab by the Japanese regulatory authority, this post-marketing observational study (PMOS) was conducted. The study investigated the long-term safety of adalimumab, particularly associated with the development of infections and malignant tumors. Data was collected once every 6 months up to 3 years.

ELIGIBILITY:
Inclusion criteria:

1. Participants who received adalimumab in accordance with its indications for treatment and dosage regimens.
2. Participants who used adalimumab continuously.
3. Participants without current or past history of malignant tumors.
4. Participants evaluated for Disease Activity Score 28 - 4 Erythrocyte Sedimentation Rate (DAS28-4ESR).
5. Participants evaluated by Health Assessment Questionnaire (HAQ) or Modified Health Assessment Questionnaire (MHAQ) prior to the initiation of adalimumab treatment in the all-case PMOS.

Exclusion criteria:

1. Contraindications according to the package insert.
2. Participants with serious infections.
3. Participants with tuberculosis.
4. Participants with a history of hypersensitivity to any ingredient of adalimumab.
5. Participants with demyelinating disease or a history of demyelinating disease.
6. Participants with congestive cardiac failure.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who received adalimumab in accordance with its indications for treatment and dosage regimens.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2009-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Kurimoto, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The primary reason for discontinuation was not collected for 224 participants listed under the category of 'multiple reasons per participant' (Insufficient effect (n=76), other reasons (n=43), economic reasons (n=2), AEs (n=41), no further visits (including change of hospital) (n=39), discontinued by the patient request (n=17), and unknown (n=8)).
Period: Overall Study
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Started | 552
Completed | 284
Not Completed | 268
Not completed — Off-Label Use of Adalimumab | 8
Not completed — Did Not Continue Use of Adalimumab | 26
Not completed — History/comorbidity of malignant tumor | 3
Not completed — Participants Without Case Report Form | 7
Not completed — Multiple Reasons Per Participant | 224

BASELINE CHARACTERISTICS:
Population: Safety analysis set, defined as participants who did not violate protocol criteria.
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Number analyzed (Participants) | 508
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 416
  Male | 92

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Drug Reactions (ADRs)
Description: An ADR was any unfavourable or unintended response (adverse event) that could possibly be related to adalimumab treatment. ADRs were assessed and data are presented as percentage of participants.
Time Frame: From the initiation of adalimumab treatment, every 6 months up to 3 years.
Population: Safety analysis set, defined as participants who did not violate protocol criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Number analyzed (Participants) | 508
Percentage of participants | 33.3

2. Secondary Outcome: Incidence of Infections and Malignant Tumors
Description: Participants were evaluated for the presence/absence of malignant tumors and infections. Data are presented as percentage of participants.
Time Frame: From the initiation of adalimumab treatment, every 6 months up to 3 years.
Population: Safety analysis set, defined as participants who did not violate protocol criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Number analyzed (Participants) | 508
Percentage of participants
  Infections | 16.1
  Malignant Tumors | 1.2

3. Secondary Outcome: Percentage of Participants With Disease Activity Score 28 - 4 Erythrocyte Sedimentation Rate (DAS28-4ESR) < 2.6 by Visit
Description: DAS28-4ESR, a combined index that measured activity of rheumatoid arthritis, was calculated based on: (1) the number of tender joints among 28 joints evaluated; (2) the number of swollen joints among 28 joints evaluated; (3) general health evaluated by a visual analog scale (VAS); and (4) ESR. DAS28-4ESR scores ranged from 0 (no disease activity) to 10 (maximal disease activity); decrease in DAS28-4ESR scores indicate improvement of disease. DAS28-4ESR score < 2.6 was defined as clinical remission of rheumatoid arthritis. Data are presented as percentage of participants.
Time Frame: Baseline (Week 0), Week 4, Week 12, Week 24, Year 1, Year 1.5, Year 2, Year 2.5, and Year 3
Population: Efficacy analysis set, defined as safety analysis set excluding participants without evaluable DAS28-4ESR score and lack of Modified Health Assessment Questionnaire (MHAQ) data prior to drug administration.
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Number analyzed (Participants) | 429
Percentage of participants
  Baseline (Week 0) | 2.8
  Week 4 | 14.5
  Week 12 | 20.0
  Week 24 | 29.6
  Year 1 | 33.6
  Year 1.5 | 37.1
  Year 2 | 36.6
  Year 2.5 | 38.2
  Year 3 | 36.4

4. Secondary Outcome: Percentage of Participants With Modified Health Assessment Questionnaire (MHAQ) Score ≤ 0.5 by Visit
Description: MHAQ was a participant-reported questionnaire that measured quality of life in terms of physical function of participants with rheumatic diseases. Participants assessed their ability to do each task over the past 6 months using the following response categories (score): without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score from 0 to 3, where 0 represented no disability and 3 very severe, high-dependency disability. MHAQ score ≤ 0.5 was defined as clinical remission, signifying normal physical function. Data are presented as percentage of participants.
Time Frame: Baseline (Week 0), Week 24, Year 1, Year 1.5, Year 2, Year 2.5, and Year 3
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Number analyzed (Participants) | 426
Percentage of participants
  Baseline (Week 0) | 43.4
  Week 24 | 53.5
  Year 1 | 63.6
  Year 1.5 | 63.6
  Year 2 | 66.0
  Year 2.5 | 65.7
  Year 3 | 66.2

ADVERSE EVENTS:
Time Frame: From the initiation of adalimumab treatment, every 6 months up to 3 years.
Description: The occurrence, type of adverse events, date of onset, seriousness (reasons for serious events), outcome (type of outcome and date of evaluation), measures taken regarding adalimumab and use of symptomatic treatment, causal relationship between adalimumab and adverse events, and laboratory findings were assessed.
Arm/Group | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection
Serious Adverse Events (participants affected / at risk) | 86/508
Other Adverse Events (participants affected / at risk) | 211/508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection (N=508)
Acute tonsillitis (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Epstein-Barr virus infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 2
Listeriosis (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia haemophilus (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 2
Pneumonia bacterial (Infections and infestations) | 4
Purulence (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Splenic lesion (Blood and lymphatic system disorders) | 1
Amyloidosis (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Anxiety disorder (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Vertigo (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Aortic rupture (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 1
Pyrexia (General disorders) | 1
Abasia (General disorders) | 1
Deformity (General disorders) | 1
Computerised tomogram thorax abnormal (Investigations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 5
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg/0.8 mL Syringe for Subcutaneous Injection (N=508)
Acute tonsillitis (Infections and infestations) | 1
Atypical pneumonia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 21
Bronchopneumonia (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 4
Chronic sinusitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Epstein-Barr virus infection (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 9
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Listeriosis (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Otitis media (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 10
Pneumonia haemophilus (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Pulmonary mycosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Subcutaneous abscess (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Arthritis bacterial (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 3
Pneumonia bacterial (Infections and infestations) | 4
Atypical mycobacterial infection (Infections and infestations) | 1
Purulence (Infections and infestations) | 2
Oral herpes (Infections and infestations) | 4
Tinea manuum (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 5
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Splenic lesion (Blood and lymphatic system disorders) | 1
Amyloidosis (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 2
Anxiety disorder (Psychiatric disorders) | 1
Cerebral infarction (Nervous system disorders) | 3
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyslalia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 4
Aortic rupture (Vascular disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 20
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gingival swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Parotid gland enlargement (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Chronic hepatitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 26
Liver disorder (Hepatobiliary disorders) | 5
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 4
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 10
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Neurogenic bladder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 1
Chest discomfort (General disorders) | 1
Chills (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 9
Injection site pruritus (General disorders) | 1
Injection site rash (General disorders) | 3
Injection site reaction (General disorders) | 1
Pyrexia (General disorders) | 4
Abasia (General disorders) | 1
Injection site swelling (General disorders) | 1
Deformity (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Liver function test abnormal (Investigations) | 3
Platelet count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Blood beta-D-glucan increased (Investigations) | 2
Computerised tomogram thorax abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 3
Cell marker increased (Investigations) | 3
Arthropod sting (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Frostbite (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 7
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.